CLINICAL TRIAL: NCT04578093
Title: Investigating an Implementation Strategy for a Peer-based Intervention to Prevent Teen Pregnancy
Brief Title: Implementation Strategy for a Peer-based Intervention to Prevent Teen Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI No Longer at Institution
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 20-0250
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Contraception Behavior
Keywords: teen pregnancy, adolescent contraception
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: case-control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will receive adjusts curriculum
  Interventions: Behavioral: LARC peer-based curriculum
- Control (No Intervention): Will receive unadjusted curriculum

INTERVENTIONS:
Behavioral: LARC peer-based curriculum — Peer-based educational videos and supplemental activities
  Arms: Intervention

SUMMARY:
Previously studied peer-based educational videos on LARC (long-acting reversible contraceptive) devices will be incorporated into a high school health curriculum. This will then be administered to the intervention high school. Outcomes including LARC knowledge, attitudes and uptake will be compared to a control high school.

ELIGIBILITY:
Inclusion Criteria:

female, never used LARC, attending high school, less than 20 yo

Exclusion Criteria:

used LARC

Ages: 13 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — only females can receive LARC
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Inquiries made of provider | 6 months
  Incidence of teenagers initiating LARC discussion or asking provider questions about LARC when visiting the school-based healthcare clinic provider.

SECONDARY OUTCOMES:
LARC uptake | 3 years
  Incidence of teenager using IUD or subnormal implant.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja R Patel, MD, MPH, MMS, Principal Investigator — UTMB